CLINICAL TRIAL: NCT04117451
Title: The Effect of Propolis Mouthwash Compared to Chlorhexidine Mouthwash on Oral and Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Raul Bescos, Principal investigator, University of Plymouth
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UPlymouth
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Blood Pressure; Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Propolis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine (Sham Comparator): Chlorhexidine mouthwash will be provided to participants for a week to rinse the mouth twice a day.
  Interventions: Other: Propolis
- Propolis (Experimental): Propolis mouthwash will be provided to participants for a week to rinse the mouth twice a day.
  Interventions: Other: Propolis

INTERVENTIONS:
Other: Propolis — Investigating the impact of propolis mouthwash on oral and cardiovascular health

SUMMARY:
The oral microbiome has recently emerged as a key contributor in nitric oxide (NO) homeostasis and vascular control by increasing nitrite bioavailability. Antibacterial mouthwash containing chlorhexidine has been shown to be effective in inhibiting the nitrate-reducing activity of oral bacteria, and increasing blood pressure in normotensive and hypertensive individuals. Recent research has also shown that chlorhexidine mouthwash lowered salivary pH and increased salivary lactate and glucose. This was also associated with changes on the activity and diversity of oral bacteria that are susceptible to increase the risk of periodontal disease. On the other hand, mouthwash containing propolis has similar antimicrobial effects than chlorhexidine, but adding some positive outcomes such as increased salivary antioxidant capacity. This may suggest that propolis mouthwash modulates the activity/diversity of oral bacteria. Thus, this study aims to investigate the effect of propolis mouthwash on the nitrate-reducing activity of oral bacteria and vascular function compared to chlorhexidine in healthy humans.

DETAILED DESCRIPTION:
Methods:

Participants: Adult healthy and non-smoker individuals will be recruited. The study will be approved by the Human Ethics Committee of the University of Plymouth.

Main protocol: Participants will visit the laboratory on two different occasions. At the first visit, basic anthropometrical measurements will be taken before to collect a blood (6 mL) and saliva (3 mL) samples under fasting conditions. Then, the nitrate reducing capacity of oral bacteria will be measured using a 10 mL of a free-nitrite water solution containing sodium nitrate. Participants will rinse their mouth for 5 min. Then, the mouth rinse will be collected into a sterile tube to analyse the absolute concentration of nitrite. Following this, blood pressure will be taken in triplicate on the left arm using an electronic sphygmomanometer. Then, microvascular function will be measured on the left forearm (extensor digitorum) using a hyperaemia reactive test. At the end of this visit and following a double-blind and non-cross over design participants will be allocated in one group: 1) chlorhexidine mouthwash or 2) propolis mouthwash. Participants will be given 14 tubes of 10 mL of mouthwash to rinse their mouth twice a day for a week before to return to the laboratory a week later and to undertake the same measurements.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals between 18 and 50 years old

Exclusion Criteria:

1. Smoking
2. To have hypertension, dyslipidaemia, diabetes, cancer or other physiological and mental disorders
3. Existing interventions affecting the oral bacteria: mouthwash, tongue scrapes
4. To have taken antibiotics within the last month.
5. In females, to have irregular menstrual periods, less than or greater than 28 days over the last 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Enhanced activity of oral bacteria | 1 week
  The nitrate-reducing nitrate activity of oral bacterial will be measured before and after each treatment
Enhanced cardiovascular function | 1 week
  Blood pressure and microvascular response to a hyperaemia reactive test will be measured before and after each treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Plymouth, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared for collaborative research.